

#### **Informed Consent**

Medical Record Number

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

A Phase II Trial of Cetuximab for Patients with Advanced or Metastatic Chordoma

| 2020-0217 |
|-------------------------------------------------------------------------|
| Subtitle: Cetuximab for Advanced/Metastatic Chordoma_ICD ver. 11Dec2024 |
| Study Chair: Anthony P. Conley, MD |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

Participant's Name

The goal of this clinical research study is to learn the effectiveness and safety of cetuximab in patients with advanced or metastatic (has spread) chordoma.

**This is an investigational study.** Cetuximab is FDA approved and commercially available for the treatment of many types of cancer. It is not approved for treatment of advanced or metastatic chordoma.

The study drug may help control the disease. Future patients may benefit from what is learned from this study. There may be benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. You may not want to take part in this study due to the potential for long stays out of town as needed for study visits.

You can read a full list of potential side effects below in the Possible Risks section of this consent.

You may continue taking cetuximab for as long as the study doctor thinks it is in your best interest.

Cetuximab will be provided at no cost to you while you are on study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive surgery and/or radiation therapy if indicated. You may choose to receive non-standard chemotherapies. You may choose to receive other investigational therapy, if available. The study doctor will discuss with you the possible risks and benefits of these treatments. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

#### 1. STUDY DETAILS

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will help the doctor decide if you are eligible. If you have had some these tests recently, they may not need to be repeated.

- You will have a physical exam.
- You will have a triplicate EKG (3 EKGs in a row) to check your heart function.
- Blood (up to 3 tablespoons) will be drawn for routine tests. This blood will also be used to test for HIV and hepatitis. If you test positive for HIV, you cannot take part in this study. If you have hepatitis, you may still be eligible.
- Urine will be collected for routine tests.
- You will have an MRI, CT scan, and/or PET/CT scan to check the status of the disease.
- Leftover tumor tissue from a previously performed procedure will be collected to check your genetic mutation (change) status and for biomarker testing.
   Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug. If no leftover tissue is available, you will have tumor biopsy. To collect a tumor tissue biopsy, the affected area is numbed with anesthetic and a small amount of tissue is removed. The study doctor will tell you if an additional biopsy is needed.
- If you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

Up to 29 participants will be enrolled in this study. All will take part at MD Anderson.

#### **Study Drug Administration**

If you are eligible to take part in this study, you will receive cetuximab by vein 1 time every 2 weeks while you are on study (Days 1 and 15 of each 28-day study cycle). The dose will be given over about 2 hours.

You will no longer be able to receive cetuximab if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits described below.

#### **Study Visits**

# On Day 1 of Cycle 1:

- You will have a physical exam.
- Blood (up to 2 tablespoons) will be drawn for routine tests.
- Blood (about 1 teaspoon) will be drawn for biomarker testing.
- You will complete a questionnaire about any symptoms you are having that may be caused by the disease. The questionnaire should take about 15 minutes to complete.
- If you can become pregnant, urine will be collected for a pregnancy test.

## On Day 1 of Cycle 2:

- You will have a physical exam.
- Blood (up to 2 tablespoons) will be drawn for routine tests.
- If you are able to become pregnant, urine will be collected for a pregnancy test.

At some point during Week 8 (at the end of Cycle 2 or beginning of Cycle 3), you will have a tumor biopsy and blood (about 1 teaspoon) drawn for biomarker testing.

At the end of every 2 cycles (Cycles 2, 4, 6, and so on), you will have an MRI, CT scan, and/or PET-CT scan to check the status of the disease.

## On Day 1 of Cycles 3:

- You will have a physical exam.
- Blood (up to 2 tablespoons) will be drawn for routine tests.
- You will complete the symptom questionnaire.
- If you can become pregnant, urine will be collected for a pregnancy test.

## On **Day 1** of **Cycles 4** and beyond:

- You will have a physical exam.
- Blood (up to 2 tablespoons) will be drawn for routine tests.
- If you are able to become pregnant, urine will be collected for a pregnancy test.

### **Follow-Up Visit**

About 4 to 6 weeks after you stop receiving cetuximab:

- You will have a physical exam.
- Blood (up to 2 tablespoons) will be drawn for routine testing.

## **Long-Term Follow Up**

You will be contacted (in person or by telephone) every 3 months for about 2 years. You will be asked about your health. If you are contacted by phone, each call should take about 10 minutes. The study staff may also follow up by contacting a family member if you choose to provide a family member's contact information, contacting another treating physician, or by reviewing your public health records.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the treatment/procedures.

## **Cetuximab Side Effects**

# Common (occurring in more than 20% of patients)

| <ul> <li>fatigue/lack of energy</li> <li>headache</li> <li>difficulty sleeping</li> <li>fever</li> <li>skin rash (possibly acnelike), peeling, and/or itching</li> <li>dry skin</li> <li>nail changes</li> <li>low blood levels of magnesium (possible weakness, muscle cramps and/or irregular heartbeat)</li> <li>weight loss</li> <li>dehydration</li> </ul> | <ul> <li>constipation</li> <li>diarrhea</li> <li>mouth blisters/sores (possible difficulty swallowing)</li> <li>vomiting</li> <li>nausea</li> <li>abnormal liver tests (possible liver damage)</li> <li>weakness</li> </ul> | <ul> <li>pain</li> <li>nerve damage (loss of sensory function)</li> <li>difficulty breathing</li> <li>cough</li> <li>sore throat</li> <li>infection</li> <li>severe rash at the site of previous radiation</li> </ul> |
|---|---|---|
|---|---|---|

Cetuximab may cause an increased risk of infection, such as pneumonia. This infection may occur anywhere. It may become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# Occasional (occurring in 3-20% of patients)

| • confusion | dry mouth | immune reaction |
|---|---|---|
| <ul> <li>depression</li> </ul> | <ul> <li>abnormal taste</li> </ul> | <ul> <li>infusion reaction</li> </ul> |
| <ul><li>anxiety</li></ul> | <ul> <li>upset stomach</li> </ul> | (possible chills and/or |
| <ul> <li>chills/shivering</li> </ul> | <ul><li>joint pain</li></ul> | hives) |
| • | <ul><li>bone pain</li></ul> | |

# Rare but serious (occurring in fewer than 3% of patients)

| <ul> <li>inflammation of the<br/>membranes around the<br/>spinal cord and brain<br/>(possible headache and/or<br/>coma)</li> </ul> | very severe blistering<br>skin disease (loss of<br>large portion of skin<br>and/or ulcers of the<br>skin and digestive<br>tract) | <ul> <li>large skin blisters</li> <li>lung inflammation<br/>(possible difficulty<br/>breathing)</li> </ul> |
|---|---|---|
|---|---|---|

# **Other Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

During the **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

**CT scans** send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

A **PET scan** may cause you to feel "closed in" while lying in the scanner. However, the scanner is open at both ends and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or technicians will give comfort, or the scanning will be stopped.

The PET scan exposes your body to radiation. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.

The type of **biomarker testing and genetic testing** being performed in this study will not provide you or your doctor information about diseases that are passed down in families. It will not tell the study researchers anything that will prevent you from getting health insurance, and it will not tell the study researchers anything about any diseases or conditions you may get in the future.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

This study may involve unpredictable risks to the participants.

## **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Birth Control Specifications: If you can become pregnant or father a child, you must use 2 highly effective methods of birth control while you are on study and for at least 90 days after your last dose of study drug. Highly effective methods of birth control are those that, alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly and include:

- Birth control pills, insertions, injections or implants, as long as you remain on the same treatment throughout the entire study and have been using this method for enough period of time to ensure it is effective
- Copper-containing intrauterine device (IUD)
- Male condom or female condom used with a spermicide (foam, gel, film, cream, or suppository)
- Male sterilization with confirmed absence of sperm in the post-vasectomy ejaculate
- Bilateral tubal ligation ("tubes tied") or bilateral salpingectomy (removal of both Fallopian tubes)

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or Eli Lilly for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result

from your participation in this research.

You will receive no compensation for taking part in this study.

## **Additional Information**

- 4. You may ask the study chair (Dr. Anthony Conley, at 713-796-3626) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. The study staff may ask if they can continue collecting the results of routine care from your medical record. If you agree, this data will be handled the same as research data.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Eli Lilly, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: Eli Lilly.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

#### **Future Research**

Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and Eli Lilly, and/or shared with other researchers and/or institutions for use in future research.

## **Samples**

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research. Leftover samples stored by Eli Lilly will be used in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

#### **Genetic Research**

Samples collected from you as part of this study will be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you. The same level of data protection that covers your individual data does not apply to summary results (when data from the whole study is combined).

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most

employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

# <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Eli Lilly, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will do its best to protect the privacy of your records, but it is possible that once information is shared with people listed on this form, it may be released to others. If this happens, your information may no longer be protected by federal law.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD

Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.

E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# CONSENT/AUTHORIZATION I understand the information in this consent form. I have had a chance to read the

| consent form for this study, or have had it read to me. I have about it, ask questions, and talk about it with others as nee permission to enroll me on this study. By signing this cons any of my legal rights. I will be given a signed copy of this | eded. I give the study chair<br>sent form, I am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT | |
| I was present during the explanation of the research to be | performed under this protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY A witness signature is only required for non-English speakers utilizing short form consent process (VTPS) and patients who are illiterate. | CHAIR) |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSE | ENT |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant ar representative, using language that is understandable and have fully informed this participant of the nature of this student and risks and that the participant understood this explanation | appropriate. I believe that I dy and its possible benefits |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |